CLINICAL TRIAL: NCT04678921
Title: A Phase 1 Study of TJ210001 Administered in Subjects With Relapsed or Refractory Advanced Solid Tumors
Brief Title: Study of TJ210001 Administered in Subjects With Relapsed or Refractory Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: I-Mab Biopharma US Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TJ210001STM101
Record Dates: First submitted 2020-12-15; First posted 2020-12-22 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Solid Tumor; Metastatic Cancer; Advanced Cancer
Keywords: monoclonal antibody; anti-C2aR
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose Level 1 (Experimental): 1mg/kg Q1W
  Interventions: Drug: TJ210001
- Dose Level 2 (Experimental): 3 mg/kg Q1W
  Interventions: Drug: TJ210001
- Dose Level 3 (Experimental): 10mg/kg Q1W
  Interventions: Drug: TJ210001
- Dose Level 4 (Experimental): 15 mg/kg Q1W
  Interventions: Drug: TJ210001

INTERVENTIONS:
Drug: TJ210001 — human anti-C5aR monoclonal antibody
  Other Names: MOR210; MOR044254; WBP2191

SUMMARY:
This is an open label, multi-center, multiple dose Phase 1 study to evaluate the safety, tolerability, MTD or MAD, PK, and PD of TJ210001 in subjects with relapsed or refractory advanced solid tumors. Beginning with Dose Level 1, TJ210001 will be given every week starting on Cycle 1 Day 1 (C1D1). The criteria for dose escalation/de-escalation will be based on the Bayesian optimal interval (BOIN) design with sequentially enrolled cohorts. The BOIN design is implemented in a simple way similar to the traditional 3+3 design but is more flexible and possesses superior operating characteristics that are comparable to those of the more complex model-based designs, such as the continual reassessment method (CRM).

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, of any race, age ≥ 18 years;
2. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1;
3. Willingness and ability to consent for self to participate in study and the ability to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures;
4. Histologically confirmed advanced or metastatic cancer in patients who are refractory to or intolerant to all available therapy. Patients who received prior PD-1/PD-L1 checkpoint inhibitor or prior CTLA-4 inhibitor therapy may enroll if they did not experience Grade 3 immune-related toxicity (exceptions may be allowed provided these toxicities have resolved e.g. Grade 3 endocrinopathy that is resolved or clinically stable with hormone replacement therapy). There is no limit to the number of prior treatment regimens;
5. At least one measurable lesion as defined by RECIST 1.1;
6. Resolution of all acute adverse events resulting from prior cancer therapies to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v5.0 Grade ≤ 1 or baseline (except alopecia or neuropathy);
7. Considered by the Investigator to be an appropriate candidate for a Phase 1 clinical study, with a life expectancy of ≥ 12 weeks;
8. Adequate organ function as defined by the following criteria:

   1. Absolute neutrophil count (ANC) ≥ 1500/μL (≥1.5 × 109/L) without growth factor support for 7 days (14 days if on pegfilgrastim) prior to study treatment;
   2. Platelets ≥ 100,000/μL (≥ 100 ×109/L) without transfusion support within 14 days prior to study treatment;
   3. Hemoglobin ≥ 9.0 g/dL without transfusion support within 14 days prior to study drug administration (erythropoietin or darbepoetin permitted);
   4. Adequate renal function and serum creatinine ≤ 1.5 times the ULN or estimated creatinine clearance ≥ 30 mL/min by Cockcroft-Gault equation4;
   5. Total serum bilirubin ≤ 1.5 times the ULN, unless patient has documented Gilbert's disease in which case bilirubin ≤ 3.0 times the ULN;
   6. Serum aspartate transaminase (AST; serum glutamic oxaloacetic transaminase [SGOT]) and serum alanine transaminase (ALT; serum glutamic pyruvic transaminase [SGPT]) ≤ 2.5 times upper limit of normal (ULN) or ≤ 5 times ULN in cases of liver metastases
   7. Albumin ≥ 3.0 g/dL;
   8. Prothrombin Time (PT) ≤ 1.5 times the ULN, or 11 to 15 seconds in the absence of a normal range; partial thromboplastin time (PTT) or activated partial thromboplastin time (aPTT) ≤ 1.5 times the ULN; and international normalized ratio (INR) ≤ 1.5 times the ULN unless the subject is receiving anticoagulant therapy.
9. Subject with a QT interval corrected for heart rate using Fridericia's formula (QTcF) and/or QT interval corrected for heart rate using Bazett's formula of < 470 msec for both males and females;
10. A 28-day washout period after the completion of programmed death-1 (PD-1)/PD-L1 therapy;
11. Women of childbearing potential (WOCBP) must:

    1. Agree to use at least 2 effective contraceptive methods (1 highly effective method in combination with a barrier method; oral, injectable, or implantable hormonal contraceptive; tubal ligation; intra-uterine device; barrier contraceptive with spermicide; or vasectomized partner), one of which must be barrier, from signing the ICF, throughout the study, and for up to 12 weeks following the last dose of TJ210001;
    2. Have a negative serum pregnancy test (sensitive of at least 25 mIU/ml) at screening; and have a negative serum or urine pregnancy test (Investigator's discretion) within 72 hours prior to Cycle 1 Day -1 of study treatment (note that the screening serum pregnancy test can be used as the test prior to Day -1 study treatment if it is performed within the prior 72 hours);
    3. Avoid conceiving for 12 weeks after the last dose of TJ210001;
    4. Avoid donation of ova from signing the ICF until 12 weeks after the last dose of TJ210001;
    5. Agree to ongoing urine pregnancy testing, if clinically indicated, during the course of the study.
12. Males must agree to use a condom (a latex condom is recommended) during sexual contact with a pregnant female or a female of childbearing potential and will avoid donation of sperm or having a female partner conceive from the time of signing the ICF, while participating in the study, during dose interruptions, and for at least 12 weeks after the last dose of study treatment, even if he has undergone a successful vasectomy.

Exclusion Criteria:

1. Has an active autoimmune disease requiring systemic treatment within the past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is permitted;
2. Current treatment on another therapeutic clinical trial;
3. Receipt of systemic anticancer therapy, including investigational agents, within 28 days prior to study treatment (Note: if anticancer therapy was given within 28 days prior to starting study treatment, patients are not excluded if ≥ 5 times the elimination half-life of the drug has elapsed.);
4. Prior treatment with C5aR inhibitors;
5. Prior T-cell or NK-cell therapy;
6. Major surgical procedure or significant traumatic injury within 4 weeks prior to study treatment, and must have fully recovered from any such procedure; and no date of surgery (if applicable) or anticipated need for a major surgical procedure planned within the next 6 months (The following are not considered to be major procedures and are permitted up to 14 days prior to study treatment: thoracentesis, paracentesis, port placement, laparoscopy, thoracoscopy, tube thoracostomy, bronchoscopy, endoscopic ultrasonographic procedures, mediastinoscopy, incisional biopsies, and routine dental procedures. Core biopsy and skin biopsy do not require a waiting period prior to dosing.);
7. Chest radiotherapy ≤ 28 days, wide field radiotherapy ≤ 28 days (defined as > 50% of volume of pelvic bones or equivalent), or limited field radiation for palliation ≤ 14 days prior to study treatment - such patients must have recovered adequately from any side effects of such therapy;
8. Hypertension defined as blood pressure (BP) systolic > 150 or diastolic > 90 mm Hg (Note: Initiation or adjustment of antihypertensive medication prior to study dosing is allowed provided that the average of the three most recent BP readings prior to study enrollment is ≤ 150/90 mm Hg.);
9. Ascites, pericardial or pleural effusions that required intervention within 1 month prior to study treatment;
10. Has known active CNS metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are radiologically stable, i.e., without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment;
11. Any of the following in the previous 6 months: severe/unstable angina, myocardial infarction (MI), symptomatic congestive heart failure, cerebrovascular accident, transient ischemic attack (TIA), arterial embolism, pulmonary embolism, percutaneous transluminal coronary angioplasty (PTCA), deep vein thrombosis, coronary artery bypass grafting (CABG), or New York Heart Association (NYHA) Class 3 or 4 congestive heart failure;
12. Has a diagnosis of immunodeficiency (known active HIV, hepatitis B virus, hepatitis C virus infection) or is receiving chronic systemic steroid therapy (in dosing exceeding 10mg of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug;

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-12-17 (Actual); Primary Completion 2022-11-21 (Actual); Study Completion 2022-11-21 (Actual)

PRIMARY OUTCOMES:
Incidence and Severity of Adverse Events | 90 days post last dose
  The CTCAE criteria will be used to assess adverse events on this trial.
Maximum Tolerated Dose | 21 days
  Based on DLT Definitions

SECONDARY OUTCOMES:
Pharmacokinetic Profile | 90 days post last dose
  Cmax
Pharmacokinetic Profile | 90 days post last dose
  AUC
Anti-drug Antibodies (ADA) | 90 days post last dose
  Incidence of anti-drug antibodies
Anti-drug Antibodies (ADA) | 90 days post last dose
  Concentration of anti-drug antibodies
Response Rate | Up to 2 years
  RECIST 1.1 will be used to assess response rate on this trial.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of Colorado Hospital - Anschutz Cancer Pavilion, Aurora, Colorado
  - Horizon Oncology Center, Lafayette, Indiana
  - Huntsman Cancer Institute, University of Utah, Salt Lake City, Utah
  - Virginia Cancer Specialists, Fairfax, Virginia